CLINICAL TRIAL: NCT00234637
Title: An Open-label Study to Evaluate the Efficacy and Safety of add-on Memantine [5-10 mg b.i.d (10-20 mg/Day)] to Rivastigmine [1.5-6 mg b.i.d. (3-12 mg/Day)] Treatment in Patients With Alzheimer's Disease Who Continued With Rivastigmine Treatment After a Previous Decline While on Donepezil or Galantamine Treatment
Brief Title: Rivastigmine Monotherapy and Combination Therapy With Memantine in Patients With Moderately Severe Alzheimer's Disease Who Failed to Benefit From Previous Cholinesterase Inhibitor Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CENA713BFR05
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease,; switch,; rivastigmine,; memantine
MeSH Terms: conditions — Alzheimer Disease | interventions — Rivastigmine; Memantine

INTERVENTIONS:
Drug: Rivastigmine, memantine

SUMMARY:
This is a prospective, multicenter, open-label study. Following screening and baseline assessments, eligible patients will be switched to rivastigmine and will enter the 16 week run-in rivastigmine treatment phase. After completion of assessments at the end of the run-in phase, patients who were not sufficiently stabilized on rivastigmine alone will receive add-on memantine to their rivastigmine treatment; patients who were stabilized on rivastigmine alone will have completed and be discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who have probable Alzheimer's disease according to the DSMIV criteria
* Patients treated with donepezil (5-10 mg ) or galantamine (16- 24 mg) for at least 6 months
* Patients, in the investigator's clinical judgment, not stabilized on treatment with donepezil or galantamine

Exclusion Criteria:

* Patients with evidence of severe or unstable physical illness, i.e., acute and severe asthmatic conditions, severe or unstable cardiovascular disorders, active peptic ulcer disease, hypersensitivity to cholinesterase inhibitors or memantine, clinically significant laboratory abnormalities or any patient with a medical condition which would prohibit them from completing the clinical trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2003-11; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
The proportion of responders (cognitive function stable or improved) at the end of phase 2 (vs. end of phase 1).

SECONDARY OUTCOMES:
Change in cognition at weeks 16 and 28 (end of period 1) compared to baseline
Change in caregiver burden at weeks 16 and 28 (end of period 1) compared to baseline
Change in behavior at weeks 16 and 28 (end of period 1) compared to baseline
Change in executive function at weeks 16 and 28 (end of period 1) compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Dantoine, Principal Investigator — Centre Hospitalier Universitaire
Locations (1):
- Département de Gérontologie Clinique, Limoges, Cedex, France